CLINICAL TRIAL: NCT05854147
Title: Comparison of Effects of Treadmill Training With and Without Visual and Auditory Cues for Freezing & Gait in Patients With Parkinson's Disease
Brief Title: Comparison of Effects of TT With and Without Visual and Auditory Cues for Freezing & Gait Patients With PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/534
Record Dates: First submitted 2023-03-18; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill Training With Visual and Auditory Cues (Experimental)
  Interventions: Diagnostic Test: Treadmill Training With Visual and Auditory Cues
- Treadmill Training Without Visual and Auditory Cues (Other)
  Interventions: Diagnostic Test: Treadmill Training Without Visual and Auditory Cues

INTERVENTIONS:
Diagnostic Test: Treadmill Training With Visual and Auditory Cues — Comparison of Effects of Treadmill Training With Visual and Auditory Cues
  Arms: Treadmill Training With Visual and Auditory Cues
Diagnostic Test: Treadmill Training Without Visual and Auditory Cues — Comparison of Effects of Treadmill Training Without Visual and Auditory Cues
  Arms: Treadmill Training Without Visual and Auditory Cues

SUMMARY:
To determine the comparison of effects of treadmill training with and without visual and auditory cues for freezing and gait in patients with Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

* Patient who are clinically diagnosed with Parkinson Disease. Patients from both genders. Patients with age between 45 years and above. Patient with sufficient visual and auditory capacity to receive given cues will be included

Exclusion Criteria:

* Patients with the history of neurological deficit other than PD. Patients who need assistance for walking will be excluded. Patient with any peripheral vascular disease will be excluded. Patient with history of lower limb fracture.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Mini Mental Examination Scale MME | 6 Months.
  MMS examination for Freezing and Gait in Patients With Parkinson's Disease

CONTACTS AND LOCATIONS:
Locations (1):
- Shadman Medical Care, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No